CLINICAL TRIAL: NCT03862222
Title: Atlas of Retinal Imaging in Alzheimer's Study
Acronym: ARIAS
Status: Completed | Type: Observational
Sponsor: University of Rhode Island (Other)
Collaborators: BayCare Health System (Other)
Responsible Party: Principal Investigator, Jessica Alber, Associate Professor of Neuroscience, University of Rhode Island
Other Study IDs: 900-403-2
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Mild Dementia; Aging; Cognitive Change
Keywords: retina; Alzheimer; cognitive aging; biomarker; preclinical Alzheimer's disease; ophthalmology; neurology
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Contrast Sensitivity; Blood Specimen Collection; Actigraphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood draw for proteomic, biomarker, and future genome wide association study (GWAS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cognitively normal - low risk: Adults aged 55-80 without subjective memory complaints, family history of Alzheimer's disease, or genetic risk for Alzheimer's disease.
  Interventions: Other: Retinal Imaging; Other: Pupillometry; Other: Contrast Sensitivity; Diagnostic Test: Neuropsychological Evaluation; Genetic: APOE genotyping; Other: blood draw; Other: Gait Assessment; Other: Actigraphy
- Cognitively normal - high risk: Adults aged 55-80 with subjective memory complaints, first degree family history of Alzheimer's disease, and at least one copy of the APOE E4 gene, a risk gene for Alzheimer's disease
  Interventions: Other: Retinal Imaging; Other: Pupillometry; Other: Contrast Sensitivity; Diagnostic Test: Neuropsychological Evaluation; Genetic: APOE genotyping; Other: blood draw; Other: Gait Assessment; Other: Actigraphy
- mild cognitive impairment: Adults aged 55-80 who have a confirmed diagnosis of mild cognitive impairment.
  Interventions: Other: Retinal Imaging; Other: Pupillometry; Other: Contrast Sensitivity; Diagnostic Test: Neuropsychological Evaluation; Genetic: APOE genotyping; Other: blood draw; Other: Gait Assessment; Other: Actigraphy
- mild dementia: Adults aged 55-80 with mild dementia due to probable Alzheimer's disease.
  Interventions: Other: Retinal Imaging; Other: Pupillometry; Other: Contrast Sensitivity; Diagnostic Test: Neuropsychological Evaluation; Genetic: APOE genotyping; Other: blood draw; Other: Gait Assessment; Other: Actigraphy

INTERVENTIONS:
Other: Retinal Imaging — Retinal imaging will be conducted on the Heidelberg SPECTRALIS (FDA 510k cleared) device, routinely used in clinical care in ophthalmology. Optical Coherence Tomography (OCT) and Angiography (OCT-A) sequences will be conducted, as well as a sequence examining macular pigment (MPOD).
Other: Pupillometry — Participants will complete a task studying pupillary response to light
Other: Contrast Sensitivity — Participants will complete a task evaluating contrast sensitivity
Diagnostic Test: Neuropsychological Evaluation — Neuropsychological evaluation will be completed, including testing in domains of memory, executive function, visuospatial ability, language, processing speed. Results will be used for research purposes only.
Genetic: APOE genotyping — APOE genotyping will be completed during screening to assign participants to the correct group. Results will not be shared with participants as part of the study.
Other: blood draw — Blood will be drawn and banked for proteomic, biomarker, and GWAS analysis
Other: Gait Assessment — Gait assessment will be conducted by trained researcher
  Other Names: Timed Up and Go, Timed Up and Go - Dual Task (TUG, TUG-DT)
Other: Actigraphy — Actigraphy monitors will be worn by all participants for 2 weeks after each visit to examine physical activity, movement, and sleep patterns.

SUMMARY:
The Atlas of Retinal Imaging in Alzheimer's (ARIAS) study is a 5-year study examining the natural history of retinal imaging biomarkers associated with disease risk, disease burden, and disease progression in Alzheimer's disease (AD). The objective of this project is to create a 'gold standard' reference database of structural anatomic and functional imaging of the retina, in order to enable the identification and development of both sensitive and reliable markers of AD risk and/or progression. Our ultimate goal is to develop a new screening protocol that identifies changes related to AD 10-20 years before AD is clinically visible.

DETAILED DESCRIPTION:
This will be a longitudinal, within-participants prospective natural history study. Participants will be recruited on the basis of serial referrals to the memory disorders centers at all three investigative sites, as well as by Institutional Review Board (IRB)-approved radio, social media and print advertisements. All participants will meet inclusion/exclusion criteria for one of the four (4) participant groups. All participants will be recruited into the study over a 24-month enrollment period. Once enrollment closes, participants will be followed for 3 years, with examinations at one of the four study locations at baseline, 12 months post-enrollment, 24 months post-enrollment, and 36 months post-enrollment. All exam and testing procedures are described below. All retinal imaging will be completed on an FDA-approved clinical OCT imaging system by trained study personnel (with quality assurance and participant safety managed by two Co-Principal Investigator (PI)'s and their staff). Pupillometry and contrast sensitivity vision testing will rely on FDA-approved and commercially widely available devices and standard clinical procedures. All techniques are well-known to both PI's, and these techniques have been in regular use by their clinical research and/or clinical care groups for the past 6+ years.

During the screening visit a cheek swab will be obtained to determine apolipoprotein (APOE) genotype. Enrollment and group assignment will be established once the genotyping results are received (i.e., approximately 55 minutes following cheek swab, and by the end of each screening visit), at which point individuals who meet enrollment criteria will be scheduled for their baseline visit. PIs may choose to include disclosure of APOE genotyping results in their location-specific protocol, if they have the appropriate clinical resources and local IRB approval for disclosure procedures. Genotyping results will not be released to participants or their physicians except through the process of an IRB approved, site-specific protocol for disclosure.

At each study visit (i.e., baseline, 12 months, 24 months, and 36 months) participants will undergo an eye examination and screening for ophthalmic disease, a medical screening exam, vital signs, neuropsychological assessment, a blood sample for measurement of plasma biomarkers, and a full retinal imaging exam. All participants will be asked to provide consent to allow review of medical records, including relevant imaging (including both clinical reports and Digital Imaging and Communications in Medicine (DICOM) image files for computerized tomography (CT)/ magnetic resonance imaging (MRI) and amyloid positron emission tomography (PET) neuroimaging) and cerebrospinal fluid (CSF) biomarker evidence of AD, if available. Additional clinical and experimental endpoints will include measures of gait, sleep quality, social and psychological health, and pupillometry. Assessment of sleep architecture (i.e., actigraphy measures) will be collected via wearable trackers over the course of a 2-week period following the baseline and 36-month study visits. A subset of participants, in each of the subject groups, will be asked to take an over-the-counter herbal supplement (Longvida curcumin; Verdure Sciences, Inc., www.longvida.com) for two days prior to their baseline exams.

ELIGIBILITY:
Inclusion Criteria (ALL PARTICIPANTS):

* · Individuals between the ages of 55 and 80 years old (inclusive).

  * Permitted medications stable for at least 1 month prior to screening. In particular:
  * Participants may take stable doses of antidepressants lacking significant anticholinergic side effects (if they are not currently depressed and do not have a history of major depression within the past year).
  * Adequate visual and auditory acuity to allow neuropsychological testing, as determined by the eye exam and the neuropsychologist's judgment. Hearing augmentation by hearing aids is allowed.
  * Good general health or without any clinically significant abnormalities (see exclusion criteria) that would be expected to interfere with participation in the study.
  * Participants must be willing and able to provide written informed consent.
  * Participants must have a study partner (i.e., family member, close friend, or caregiver) who can attend study appointments with them and report on their level of daily functioning.
  * As this is entirely an observational study, without treatment intervention, we will allow concurrent enrollment in other clinical trials for mild cognitive impairment (MCI) or AD, including those that involved the use of investigational drugs. Relevant information about other studies in which participants are participating (e.g., study name, sponsor) will be collected and considered as a potential statistical covariate in the statistical analysis plan (SAP).

Additional Inclusion Criteria - Healthy Control Participants

* Montreal Cognitive Assessment (MoCA) total score > 26 at screening
* Clinical Dementia Rating (CDR) 0 at screening
* An absence of substantial subjective memory complaints or worry
* No first degree relative with either diagnosed AD or suspicion of AD
* A screening genotype result showing non-carrier status for APOE ε4 allele

Additional Inclusion Criteria - High-Risk for Preclinical AD Participants

* MoCA total score > 26 at screening
* CDR 0 at screening
* No clinical diagnosis of MCI or dementia of any type
* Must have all of the following three risk factors for AD:
* Subjective memory complaints as ascertained on a standardized questionnaire (i.e., ECOG).
* A positive (suspected) first-degree family history for the disease.
* A screening genotype result showing carrier status for at least one APOE ε4 gene allele Additional Inclusion Criteria - Patients with Mild Cognitive Impairment
* MoCA total score > 19 at screening
* CDR 0.5 at screening
* A clinical diagnosis of MCI (amnestic type, but may include multiple domains) from qualified specialist or from a memory disorders clinic or center
* Score of less than or equal to 85 (1.5 SD below age and education adjusted normative data) on the RBANS Delayed Memory Index (DMI)
* Positive prior biomarker evidence of Alzheimer's disease (PET imaging or CSF study), if available

Additional Inclusion Criteria - Patients with Mild Alzheimer's Disease

* MoCA total score > 15 and < 26 at screening
* CDR 1 at screening
* A clinical diagnosis of mild AD from qualified specialist or from a memory disorders clinic or center
* Score of less than or equal to 85 (1.5 SD below age and education adjusted normative data) on the RBANS Delayed Memory Index (DMI)
* Positive prior biomarker evidence of Alzheimer's disease (PET imaging or CSF study), if available
* Informed consent provided from partner, caregiver or immediate family member, with verbal assent provided by individual patient.

Exclusion Criteria:

* · Patients with histories of other ocular or neurologic disease that could affect the results, such as unusually high refractive errors ( > or < 5.0 diopters native spherical equivalent), age related macular degeneration, diabetic retinopathy, hypertensive retinopathy, retinal vascular disease, glaucoma, optic nerve disease, cystic macular edema, large cataracts or corneal disease that may preclude visualization of the retinal fundus, substantial ocular media opacity, and/or intraocular surgery within 90 days of any study visit will be excluded.

  * History of severe brain injury or other known neurologic disease or insult, which, as described by medical records, and/or as determined by the PI's clinical judgment, has resulted in lasting cognitive sequelae that would confound the assessment and staging of potential neurodegenerative disease.
  * Geriatric Depression Scale Short Form (GDS-S 15 Items) score > 6.
  * Poorly controlled major depression or another psychiatric disorder within the past year.
  * History of alcohol or substance abuse and/or dependence within the past 2 years (DSM-V criteria).
  * History of schizophrenia or a history of psychotic features, agitation or behavioral problems within the last 3 months, which could lead to difficulty complying with the protocol.
  * Participants who, in the investigator's opinion, will not comply with study procedures.
  * Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol including:
  * History of systemic cancer within the past 5 years (non-metastatic skin cancers are acceptable).
  * History of clinically significant liver disease, coagulopathy, or vitamin K deficiency within the past 2 years.
  * History of myocardial infarction within the past six (6) months or unstable or severe cardiovascular disease including angina or congestive heart failure (CHF) with symptoms at rest.
  * History of stroke(s) with lasting impairment to vision or the visual system, coagulopathy, uncontrolled hypertension (i.e., systolic BP > 170 or diastolic BP > 100) and uncontrolled or insulin requiring diabetes. Blood pressure will be recorded on the day of each examination.
  * Evidence of enlarged ventricles and/or normal pressure hydrocephalus on review of medical records or inspection of CT/MRI of the brain based on previous clinical diagnosis (MRI) as noted in their neurological history
  * History of Parkinson's disease, Parkinsonism due to multiple system atrophy (MSA), progressive supranuclear palsy (PSP), Shy Drager Syndrome (SDS) or other neuro-degenerative dementias
  * History of symptoms of narrow-angle glaucoma (warning signs include eye pain, restricted vision, blurred vision)
  * History of elevated intraocular pressure, or medical record evidence of intraocular pressure > 20 mm Hg
  * Regular (daily) use of narcotics or antipsychotic medications.
  * New use of anti-Parkinsonian medications (e.g., sinemet, amantaine, bromocriptine, pergolide and selegiline) within 2 months prior to screening.
  * New use of anti-convulsants (e.g., phenytoin, phenobarbital, carbamazepine) within 2 months prior to screening.
  * New use of centrally active beta-blockers, narcotics, methyldopa and clonidine within 4 weeks prior to screening.
  * New use of neuroleptics or narcotic analgesics within 4 weeks prior to screening.
  * New and chronic use of long-acting benzodiazepines or barbiturates within 4 weeks prior to screening.
  * Use of short-acting anxiolytics or sedative-hypnotics more frequently than 2 times per week within 4 weeks prior to screening (note: sedative agents should not be used within 72 hours of the baseline and follow-up visits).
  * Initiation or change in dose of an antidepressant lacking significant cholinergic side effects within the 4 weeks prior to screening (use of stable doses of antidepressants for at least 4 weeks prior to screening is acceptable)
  * An anticholinergic burden score of >3 on the Anticholinergic Cognitive Burden Scale (see appendix item 9.19).
  * Known hypersensitivity to anticholinergic medications, including tropicamide eye drops.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be serial referrals from public outreach (community sample) and memory clinics, male or female, between the ages of 55-80. The cognitively normal - low risk (healthy control group) will be comprised of 25 individuals aged 55-65 and 25 individuals aged 65-80. Recruitment will take place at 3 active sites: Butler Hospital (Providence, RI), Morton Plant Hospital (Tampa, FLA) and St. Anthony's Hospital (St. Petersburg, FLA).
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Structural retinal biomarkers assessed with OCT | 5 years
  retinal nerve fiber layer (RNFL) thickness
Structural retinal biomarkers assessed with OCT | 5 years
  RNFL volume
Metabolic retinal biomarkers assessed with OCT | 5 years
  volume of retinal inclusion bodies containing beta amyloid
Metabolic retinal biomarkers assessed with OCT | 5 years
  surface area of retinal inclusion bodies containing beta amyloid
Metabolic retinal biomarkers assessed with OCT | 5 years
  macular pigment optical density (MPOD)
vascular retinal biomarkers assessed with OCT-A | 5 years
  vessel caliber
vascular retinal biomarkers assessed with OCT-A | 5 years
  vessel density
vascular retinal biomarkers assessed with OCT-A | 5 years
  area of foveal avascular zone
vascular retinal biomarkers assessed with OCT-A | 5 years
  fractal dimension
vascular retinal biomarkers assessed with OCT-A | 5 years
  area of blood flow
vascular retinal biomarkers assessed with OCT-A | 5 years
  area of blood non-flow

SECONDARY OUTCOMES:
general cognition | 5 years
  Montreal Cognitive Assessment (MoCA)
general cognition | 5 years
  Repeatable Battery for the Assessment of Neuropsychological Status - Update (RBANS-U)
processing speed, attention | 5 years
  Digit Symbol Substitution Task (DSST)
language | 5 years
  Redden Lab Speech/Language Task
memory | 5 years
  Free and Cued Selective Reminder Task (FCSRT)
physiological | 5 years
  blood proteomics - 21 protein panel
physiological | 5 years
  blood biomarkers (amyloid) measured with single molecule assay
physiological | 5 years
  blood biomarkers (phosphorylated tau) measured with single molecule assay
physiological | 5 years
  gait assessment (timed get up and go + timed get up and go dual task)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Sinoff, MD, Principal Investigator — BayCare Health System; Peter J Snyder, PhD, Principal Investigator — University of Rhode Island
Locations (4):
- United States (4):
  - Morton Plant Hospital, Clearwater, Florida
  - St. Anthony's Hospital, St. Petersburg, Florida
  - University of Rhode Island, Kingston, Rhode Island
  - Butler Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided
Plan to make retinal atlas publicly available along with study data and retinal images.